CLINICAL TRIAL: NCT03490968
Title: The Impact of Branched-Chain Amino Acid Metabolism on Limb Dysfunction in PAD (MicroPAD)
Brief Title: The Impact of Branched-Chain Amino Acid Metabolism on Limb Dysfunction in PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Joshua Beckman, Professor, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 180441; 18SFRN33900069 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2018-03-30; First posted 2018-04-06 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Subjects (Other)
  Interventions: Behavioral: Vascular Assessment
- Peripheral Artery Disease (PAD) with Supervised Exercise (Experimental): Subjects will be referred for supervised exercise therapy. Subjects will have 3 visits per week for 12 weeks. Each visit will include a minimum of 30 to 40 minutes of exercise to improve ambulation with a certified trainer.
  Interventions: Behavioral: Supervised Exercise; Behavioral: Vascular Assessment
- PAD Subjects Who Undergo Revascularization of the Leg (Active Comparator): This group of subjects are receiving leg revascularization as part of standard of care.
  Interventions: Behavioral: Vascular Assessment

INTERVENTIONS:
Behavioral: Supervised Exercise — Subjects will have 3 visits per week for 12 weeks.
  Arms: Peripheral Artery Disease (PAD) with Supervised Exercise
Behavioral: Vascular Assessment — Screen: Subjects will undergo a H&P, ankle brachial index, ECG, CBC, CMP, lipid panel, HgA1C, and urinalysis. A urine pregnancy test will be performed on women of childbearing age.
  Testing Visit 1: MRI, IV in common femoral vein with phlebotomy (60 cc total) before and after sphygmomanometric cuff occlusion of lower limb, 6-minute walk test, 4-meter walk speed test, walking impairment questionnaire, and muscle biopsy.
  Supervised exercise and leg revascularization patients will return in 12 weeks and have the same study procedures as testing visit 1, plus an ankle brachial index, repeated.

SUMMARY:
Test the theory that abnormalities in the large blood vessels that deliver blood to your leg and the very small blood vessels in your leg's muscles (invisible to the eye) work together to worsen your leg function and walking.

ELIGIBILITY:
Inclusion/exclusion criteria for Healthy Subjects

Inclusion criteria

* Male or female, age ≥ 50 years old
* Non-smoker

Exclusion criteria

* Presence of peripheral artery disease
* History of a heart attack or stroke
* Diabetes
* Active cancer
* Severe renal disease (CrCl < 60)
* Severe liver disease
* Active rheumatological diseases

Inclusion/exclusion criteria for PAD Subjects

Inclusion criteria

* Male or female, age 50 years or older
* Atherosclerotic PAD, ABI ≤0.85
* Willing to comply with protocol, attend follow-up appointments, complete all study assessments, and provide informed consent
* For Aim 3, subjects will have Rutherford stage 4 or 5 disease
* For Aim 3, subjects will be undergoing revascularization as standard of care

Exclusion criteria

* Presence of a femoral, popliteal or tibial aneurysm of the index limb
* Life expectancy less than 2 years
* A vascular disease prognosis that includes an anticipated above ankle amputation on index limb within 4 weeks of index procedure
* Renal dysfunction defined as MDRD eGFR ≤ 20ml/min/173 m2 at the time of screening
* Currently on dialysis or history of a renal transplant
* Cirrhosis or active hepatitis
* A documented hypercoagulable state
* Myocardial infarction within 6 months
* Stroke within 6 months
* Nonatherosclerotic occlusive disease of the lower extremity
* Any prior infrainguinal revascularization on index limb
* Current immunosuppressive medication, chemotherapy or radiation therapy
* Inability to have an MRI
* Exercise limitation aside from that due to PAD (i.e. COPD, degenerative joint disease, etc.)
* Women who are pregnant
* Women who are nursing
* Primary indications for systemic oral anticoagulation for active arterial or venous thromboembolic disease.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
C3/C5acylcarnitine levels in healthy control subjects. | baseline
C3/C5acylcarnitine levels in PAD exercise group after 12 weeks | Change from baseline to 12 weeks
C3/C5 acylcarnitine levels in PAD surgical bypass group | Change from baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Beckman, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sullivan AE, Behroozian A, Coolbaugh C, Shardelow E, Smith EK, Wells QS, Clair DG, Aday AW, Garrard CL 3rd, Curci JA, Holder TA, Barnett JV, Freiberg MS, Crescenzi RL, Wakeham DJ, Hearon CM Jr, Donahue MJ, Beckman JA. Microvascular Function and Ambulatory Capacity in Peripheral Artery Disease. Circ Cardiovasc Interv. 2025 Oct;18(10):e015582. doi: 10.1161/CIRCINTERVENTIONS.125.015582. Epub 2025 Sep 4. PMID 40905129